CLINICAL TRIAL: NCT07219329
Title: The Feasibility of a Nurse-Initiated Weighted Blanket in Orthopedic Surgical Patients Undergoing Total Knee Arthroplasty: A Pilot Study
Brief Title: The Feasibility of a Nurse-Initiated Weighted Blanket in Orthopedic Surgical Patients Undergoing Total Knee Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-00571
Record Dates: First submitted 2025-10-20; First posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Total Knee Replacement
Keywords: anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Weighted blanket (Experimental): Participants will receive a weighted blanket in the preoperative holding room and in the Post-Anesthesia Care Unit (PACU) after surgery.
  Interventions: Device: Weighted Blanket
- Standard of care (No Intervention): Participants will receive a non-weighted blanket in the preoperative holding room prior to and in the PACU after surgery per standard of care.

INTERVENTIONS:
Device: Weighted Blanket — 5lb weighted blanket
  Arms: Weighted blanket

SUMMARY:
The purpose of this study is to explore the acceptability and feasibility of weighted blankets in total knee replacement (TKR) patients. The study also aims to measure the difference in anxiety of adult orthopedic patients in need of total knee arthroplasty surgery who receive weighted blanket before and after surgery compared to those who receive a non-weighted blanket.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and older
2. Adults undergoing elective total knee arthroplasty at NYU Langone Orthopedic Hospital.
3. Adults who are scheduled to receive spinal anesthesia.
4. Subjects with a planned same day discharge to home from the PACU

Exclusion Criteria:

1. cognitive disability that would interfere with their ability to complete the study's pre and post assessments (e.g. dementia, non-verbal)
2. subject disclosed history of pre-existing anxiety disorder, claustrophobia, epilepsy, respiratory conditions (e.g. obstructive sleep apnea (OSA), asthma), skin conditions (e.g. pressure injury), which are contradictions for weighted blanket.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Time participants used weighted blanket | PACU discharge (~1-3 hours post-surgery)
  Outcome measure assessed via investigator-created Weighted Blanket Feasibility Question in Post-Anesthesia Care Unit (PACU). Question asks "How long would you estimate that you used the weighted blanket?" Patient-reported estimate in minutes.
Number of participants who would use a weighted blanket in the future | PACU discharge (~1-3 hours post-surgery)
  Outcome measure via investigator-created Weighted Blanket Acceptability Question in PACU. The question asks the participant "If you were offered a weighted blanket in the future, would you choose to use it?" with choices of "yes", "no", and "unsure" and then asked to explain their choice.

SECONDARY OUTCOMES:
Change in short Spielberger State-Trait Anxiety Inventory (SSTAI) score | Baseline (before blanket application), PACU discharge (~1-3 hours post-surgery)
  The STAI-5 consists of 5 items relating to anxiety, each item is scored on a 4-point scale. Scores range from 5 to 20, with higher scores indicating more anxiety.
Change in Numeric Pain Rating Scale (NPRS) score | Baseline (before blanket application), PACU discharge (~1-3 hours post-surgery)
  Pain is assessed on the NPRS from 0 (No pain) to 10 (Severe pain).
Richmond Agitation-Sedation Scale (RASS) score | PACU discharge (~1-3 hours post-surgery)
  The RASS consists of a 10-point scale.. Positive scores indicate agitation, with +4 being the most severe (combative), and negative scores indicate sedation, with -5 being the deepest level of sedation (unarousable). A score of 0 indicates the patient is alert and calm.
Change in heart rate | Baseline (before blanket application), PACU discharge (~1-3 hours post-surgery)
Change in blood pressure | Baseline (before blanket application), PACU discharge (~1-3 hours post-surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Wong, MS, RN, CPAN, ONC, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Study participants did not provide consent for data sharing beyond the study team and institutional oversight. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.